CLINICAL TRIAL: NCT00015028
Title: CS1008A Efficacy/Safety Trial of Buprenorphine/Naloxone
Brief Title: Buprenorphine/Naloxone for Opiate-Dependence Treatment - 1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Collaborators: Cincinnati MDRU (Other)
Purpose: Treatment
Other Study IDs: NIDA-5-0012-1; Y01-5-0012-1
Record Dates: First submitted 2001-04-18; First posted 2001-04-18 (Estimated); Last update posted 2017-01-16 (Estimated); Status verified 1996-11

CONDITIONS: Opioid-Related Disorders; Substance-Related Disorders
Keywords: opioid dependence
MeSH Terms: conditions — Opioid-Related Disorders; Substance-Related Disorders | interventions — Buprenorphine, Naloxone Drug Combination

INTERVENTIONS:
Drug: Buprenorphine/naloxone

SUMMARY:
The purpose of this study is to determine the efficacy and safety of a buprenorphine/naloxone sublingual tablet formulation as an office-based therapy for opiate-dependence treatment. The developmental objective for this combination product is an expansion of therapeutic options for the treatment of opiate dependence.

DETAILED DESCRIPTION:
This multicenter pivotal clinical trial was comprised of two phases. The first phase, which was four weeks in length, was double-blind placebo controlled and was primarily used to evaluate the efficacy of buprenorphine/naloxone. The second phase, lasting 48 weeks, was primarily conducted to determine the safety of buprenorphine/naloxone.

ELIGIBILITY:
Inclusion Criteria:

1. DSM-IV (Diagnostic and Statistical Manual of the American Psychiatric Association) diagnosis of current opiate dependence.
2. Individuals seeking opiate-substitution pharmacotherapy for opiate dependence.
3. Males and non-pregnant, non-nursing females, 18 to 59 years of age (inclusive).
4. Individuals able to give informed consent and willing to comply with all study procedures (e.g., providing of urine samples under observation, completing questionnaires).

Exclusion Criteria:

1. Any acute or chronic medical condition that would make participation in the study medically hazardous (e.g., acute hepatitis, unstable cardiovascular, hepatic, or renal disease, unstable diabetes, symptomatic AIDS; not HIV-seropositivity alone).
2. Aspartate or alanine aminotransferase (AST, ALT) levels greater than three times the upper limit of normal.
3. Individuals currently taking systemic anti-retroviral or anti-fungal therapy.
4. Current dependence (by DSM-IV criteria) on any psychoactive substance other than opiates, caffeine, or nicotine.
5. Current, primary, Axis I psychiatric diagnosis other than opiate, caffeine, or nicotine dependence.
6. Females of childbearing potential who do not agree to use a medically acceptable method of birth control. Acceptable methods include

   1. oral contraceptive,
   2. barrier (diaphragm or condom) - a spermicide is not required due to the possibility of local irritation and allergic type reactions, but are recommended for use,
   3. levonorgestrel implant,
   4. intrauterine progesterone contraceptive system,
   5. medroxyprogesterone acetate contraceptive injection, or
   6. complete abstinence.
7. Enrollment in an opiate-substitution (i.e., methadone, levo-alpha-acetylmethadol) treatment program within 45 days of enrolling in the present study.
8. Individuals having taken (licitly or illicitly) LAAM, methadone, or naltrexone within days of enrolling in the present study.
9. Individuals having taken buprenorphine, other than as an analgesic, within 365 days of enrolling in the present study.
10. Participation in an investigational drug or device study within 45 days of enrolling in the present study.
11. Anyone, who in the opinion of site principal investigator, would not be expected to complete the first phase of the study protocol (e.g., due to pending incarceration or probable relocation from the clinic area).

Ages: 23 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0
Dates: Start 1996-11; Primary Completion 1996-12 (Actual); Study Completion 1997-01 (Actual)

PRIMARY OUTCOMES:
Craving
Drug use
HIV risk behaviors
Adverse events
Medical evaluation

CONTACTS AND LOCATIONS:
Overall Officials: Eugene Somoza, M.D., Ph.D., Principal Investigator — Cincinnati MDRU
Locations (1):
- Cincinnati MDRU, Cincinnati, Ohio, United States